CLINICAL TRIAL: NCT00000662
Title: A Treatment IND for Retrovir Brand Zidovudine (AZT) Therapy of Pediatric Patients With HIV Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Purpose: Treatment
Other Study IDs: TX 304; FDA 43A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 1992-04

CONDITIONS: HIV Infections
Keywords: Drugs, Investigational; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To facilitate the use of zidovudine (AZT) in children who are 3 months to 12 years of age who are HIV-infected and either symptomatic or have a CD4 cell count < 400 cells/mm3 and to monitor adverse effects of AZT.

Previous studies with pediatric patients have shown improvements in clinical, immunologic, and virologic parameters with administration of AZT.

DETAILED DESCRIPTION:
Previous studies with pediatric patients have shown improvements in clinical, immunologic, and virologic parameters with administration of AZT.

This Treatment IND (investigational new drug) is an open label, uncontrolled protocol. AZT is ordered and prescribed by the patient's physician. The physician is responsible for obtaining informed consent, assuring that the patient meets the eligibility criteria, dispensing the medication to the patient, monitoring the patient's condition on treatment, and reporting required data to the project coordinating center.

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed:

* Blood transfusions for hematologic toxicity.

Criteria for children 3 months to less than 15 months of age:

* Patient must be HIV antibody-positive by repeated reactive screening test (e.g., ELISA) and positive confirmatory test (e.g., Western blot).

OR

* If antibody-negative, patient must have two positive p24 antigen determinations performed at least one week apart or have had a positive HIV culture.

Patients must meet two of the following criteria:

* Be HIV culture positive or p24 antigen positive.
* Have at least one of the Class P-2 symptoms (by CDC criteria).

Be immunosuppressed defined as having:

* CD4+(T4) lymphocytes = or < 400 cells/mm3.
* Abnormal age adjusted immunoglobulin levels (IgG or IgA). Decreased helper/suppressor ratio < 1.0.

Note:

* In general, abnormal values for any of the above lab tests should be confirmed in 2 measurements at least 1 week apart, and other clinical causes for these abnormalities should be ruled out.

Criteria for children 15 months to 12 years of age:

* Patient must be HIV antibody-positive by repeated reactive screening test (e.g., ELISA) and positive confirmatory test (e.g., Western blot).

OR

* If antibody-negative, patient must have two positive p24 antigen determinations performed at least one week apart or have had a positive HIV culture.

Patients must meet one of the following criteria:

* Have at least one of the class P-2 symptoms (by CDC criteria).
* Be immunosuppressed defined as having CD4+(T4) lymphocytes = or < 400 cells/mm3, based on two measurements at least 1 week apart.

Exclusion Criteria

Co-existing Condition:

Patients with known hypersensitivity to AZT are excluded.

Patients with the following are excluded:

* Failure to meet inclusion criteria.
* Inability to obtain signed informed consent from a parent or legal guardian.
* Enrollment in another treatment protocol that expressly prohibits concomitant treatment with zidovudine (AZT).
* Enrollment in another clinical trial in which AZT is a treatment.
* Known hypersensitivity to AZT.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Primary Completion 1993-05 (Actual); Study Completion 1993-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States